CLINICAL TRIAL: NCT05508997
Title: Response of Respiratory and Hemodynamic Parameters to Positive End-Expiratory Pressure Titration for Mechanically Ventilated Obese Patients: A Randomized Clinical Trial
Brief Title: Respiratory and Hemodynamics Parameters Response to Positive End-Expiratory Pressure
Acronym: Respiratory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidy F. Ahmed (Other)
Responsible Party: Sponsor-Investigator, Heidy F. Ahmed, Doctor of physical therapy at Al kasr Al Anini teaching hospital, Cairo, Egypt, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/001827
Record Dates: First submitted 2022-08-11; First posted 2022-08-19 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Obesity Associated Disorder
Keywords: Positive end-expiratory pressure titration; Mechanical ventilator; respiratory and hemodynamics parameters; Obese patients; Reverse Trendelenburg Position.
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: group A receive Reverse Trendelenburg Position (RTP) + Positive End Expiratory Pressure (PEEP) titration, and group (B): receive Reverse Trendelenburg Position (RTP).
Who Masked: Participant, Outcomes Assessor
Masking Description: the patients were under general anesthesia didn't know which procedure they received & the outcomes assessor done by my supervisors and didn't know which result related to specific group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive End Expiatory Pressure + Reverse Trendelenburg Position (Experimental): Group A received the procedures of the physiotherapy part by applying proper positioning for better oxygenation and ventilation (Reverse Trendelenburg Position), which is the patient laid supine with the head up 30 degrees higher than the feet & received the recruitment maneuver (RM) by Positive End Expiratory Pressure (PEEP) titration
  Interventions: Device: respiratory parameters on mechanical ventilator (PEEP)
- Reverse Trendelenburg Position (Active Comparator): Group B received only the procedures of the physiotherapy part at the 3rd phase of operation by applying proper positioning for better oxygenation and ventilation (Reverse Trendelenburg Position), in which the patient laid supine with the head at 15-30 degrees higher than the feet to unload the weight of intra-abdominal contents from the diaphragm, this position:
  1. Increase pulmonary compliance, functional residual capacity (FRC), and oxygenation.
  2. Allows easier ventilation.
  3. This position called safe apnea time allows time to secure the airway before desaturation for a 20-minute positioning time.
  Interventions: Device: respiratory parameters on mechanical ventilator (PEEP)

INTERVENTIONS:
Device: respiratory parameters on mechanical ventilator (PEEP) — The 3rd & 4th phases of operation in the group (A) and (B): Each patient received one single session inside the Operation Room (OR) as one shot of the treatment procedure. Arterial Blood Gases (ABGs) were obtained to measure:
  1. Oxygenation by PaO2/FiO2 ratio with constant FiO2 = 100% (oxygen) through the procedure time as a primary outcome.
  2. Secondary outcome.
     * Ventilation by PaCO2 value from ABGs.
     * Static compliance (Cstat) was measured as the amount of recruitment of alveoli in the lung.
     * Blood pressure (systolic/diastolic) one of the hemodynamics measurements was measured pre/post the procedure in the two groups.

SUMMARY:
In this study, the sixty mechanically ventilated class I obese patients were divided into two equal groups A and B. group A received RTP position + PEEP protocol, while group B underwent RTP position protocol only. The results showed that the group A protocol has positive effects on the improvement of respiratory mechanics by significant increase the arterial oxygen partial pressure (PaO2) in mmHg to fractional inspired oxygen (FiO2), (PaO2/FiO2 ratio), partial pressure of carbon dioxide (PaCO2), and static compliance (Cstat) parameters. Moreover, a significant decrease in hemodynamics of BP& MAP was measured. While the results of the group B protocol demonstrated a non-significant increase in the PaO2/FiO2 ratio, PaCO2, and Cstat. Besides, non-significant decreases in hemodynamics of blood pressure (BP) & mean arterial blood pressure (MAP) were recorded.

DETAILED DESCRIPTION:
Objective To investigate the effect of the positive end-expiratory pressure (PEEP) titration maneuver with Reverse Trendelenburg Position (RTP) on the respiratory and hemodynamic parameters of mechanically ventilated obese patients.

Design Randomized, control trial. Participants Thirty mechanically ventilated obese patients were randomized equally as a group A to receive Reverse Trendelenburg Position (RTP) + Positive End Expiratory Pressure (PEEP) titration, and group (B): receive Reverse Trendelenburg Position (RTP).

Intervention After post-operative bariatric surgeries, the sixty mechanically ventilated obese patients immediately receive a PEEP and RTP once before the weaning through the ventilator of the operation to evaluate the response of arterial blood gases before admission to the intensive care unit ICU room.

Outcomes The primary outcomes included the respiratory parameters (PaO2/FiO2 ratio, PaCO2, Cstat), and the secondary outcomes included the hemodynamics parameters (systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial blood pressure (MAP)).

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in this study had the following criteria:

  1. Mechanically ventilated obese patients in operation room undergoing upper abdominal surgeries (bariatric) and under general anesthesia.
  2. Obese patients with BMI (30-34.9).
  3. Age 40-50 years old.
  4. Both sexes.
  5. Non-smoker.
  6. No history of disease affecting the heart & lungs.

Exclusion Criteria:

* Subjects with any of the following were excluded from the study:

  1. Severe head injury.
  2. Increase intracranial pressure and who are potentially liable to develop pathologically raised intracranial pressure.
  3. Acute pulmonary edema.
  4. Barotrauma/volutrauma.
  5. Un-drained Pneumothorax/Hemothorax.
  6. Flail chest.
  7. Low blood pressure (systolic less than 80 mmHg).
  8. Oxygen saturation is less than 90%.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Respiratory parameters | Immediately after the procedure is done in the operating room appears on the patient's monitor & patient arterial blood gases.
  The primary outcomes included the respiratory parameters partial oxygen pressure, partial carbon dioxide pressure, static compliance fractional oxygen pressure ratio

SECONDARY OUTCOMES:
Hemodynamics parameters | Immediately after the procedure is done in the operating room appears on the patient's monitor.
  The secondary outcomes included the hemodynamics parameters (SBP in mmHg, DBP in mmHg, and MAP in mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Heidy F. Ahmed, Master, Principal Investigator — Kasr al aini
Locations (1):
- Al Kasr Al Aini Teaching Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD), all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: In the next month of registration.
Access Criteria: Information will be available upon request through the following e-mail: heidy.fouad@gmail.com.

REFERENCES:
- [Background] Hibbert KA, Malhotra A. Obesity in Critically Ill Patients. In Cardiopulmonary Monitoring. 2021 (pp. 935-947). Springer, Cham. https://doi.org/10.1007/978-3-030-73387-2
- [Background] Wang QY, Ji YW, An LX, Cao L, Xue FS. Effects of individualized PEEP obtained by two different titration methods on postoperative atelectasis in obese patients: study protocol for a randomized controlled trial. Trials. 2021 Oct 15;22(1):704. doi: 10.1186/s13063-021-05671-1. PMID 34654446
- [Background] Bluth T, Teichmann R, Kiss T, Bobek I, Canet J, Cinnella G, De Baerdemaeker L, Gregoretti C, Hedenstierna G, Hemmes SN, Hiesmayr M, Hollmann MW, Jaber S, Laffey JG, Licker MJ, Markstaller K, Matot I, Muller G, Mills GH, Mulier JP, Putensen C, Rossaint R, Schmitt J, Senturk M, Serpa Neto A, Severgnini P, Sprung J, Vidal Melo MF, Wrigge H, Schultz MJ, Pelosi P, Gama de Abreu M; PROBESE investigators; PROtective VEntilation Network (PROVEnet); Clinical Trial Network of the European Society of Anaesthesiology (ESA). Protective intraoperative ventilation with higher versus lower levels of positive end-expiratory pressure in obese patients (PROBESE): study protocol for a randomized controlled trial. Trials. 2017 Apr 28;18(1):202. doi: 10.1186/s13063-017-1929-0. PMID 28454590
- [Background] Ruszkai Z, Kiss E, Laszlo I, Bokretas GP, Vizseralek D, Vamossy I, Surany E, Buzogany I, Bajory Z, Molnar Z. Effects of intraoperative positive end-expiratory pressure optimization on respiratory mechanics and the inflammatory response: a randomized controlled trial. J Clin Monit Comput. 2021 May;35(3):469-482. doi: 10.1007/s10877-020-00519-6. Epub 2020 May 9. PMID 32388650
- [Background] Silva PL, Pelosi P, Rocco PR. Ventilation in the Obese Patient. In Mechanical Ventilation from Pathophysiology to Clinical Evidence. 2022 (pp. 223-229). Springer, Cham. http://doi.org/10.1007/978-3-030-93401-9
- [Background] Bruins S, Sommerfield D, Powers N, von Ungern-Sternberg BS. Atelectasis and lung recruitment in pediatric anesthesia: An educational review. Paediatr Anaesth. 2022 Feb;32(2):321-329. doi: 10.1111/pan.14335. Epub 2021 Nov 24. PMID 34797011
- [Background] Brodsky JB. Recent advances in anesthesia of the obese patient. F1000Res. 2018 Aug 6;7:F1000 Faculty Rev-1195. doi: 10.12688/f1000research.15093.1. eCollection 2018. PMID 30135720
- [Background] De Jong A, Wrigge H, Hedenstierna G, Gattinoni L, Chiumello D, Frat JP, Ball L, Schetz M, Pickkers P, Jaber S. How to ventilate obese patients in the ICU. Intensive Care Med. 2020 Dec;46(12):2423-2435. doi: 10.1007/s00134-020-06286-x. Epub 2020 Oct 23. PMID 33095284
- [Background] Severac M, Chiali W, Severac F, Perus O, Orban JC, Iannelli A, Debs T, Gugenheim J, Raucoules-Aime M. Alveolar recruitment manoeuvre results in improved pulmonary function in obese patients undergoing bariatric surgery: a randomised trial. Anaesth Crit Care Pain Med. 2021 Jun;40(3):100775. doi: 10.1016/j.accpm.2020.09.011. Epub 2020 Nov 1. PMID 33137453
- [Background] Boone MD, Jinadasa SP, Mueller A, Shaefi S, Kasper EM, Hanafy KA, O'Gara BP, Talmor DS. The Effect of Positive End-Expiratory Pressure on Intracranial Pressure and Cerebral Hemodynamics. Neurocrit Care. 2017 Apr;26(2):174-181. doi: 10.1007/s12028-016-0328-9. PMID 27848125
- [Background] Fumagalli J, Santiago RRS, Teggia Droghi M, Zhang C, Fintelmann FJ, Troschel FM, Morais CCA, Amato MBP, Kacmarek RM, Berra L; Lung Rescue Team Investigators. Lung Recruitment in Obese Patients with Acute Respiratory Distress Syndrome. Anesthesiology. 2019 May;130(5):791-803. doi: 10.1097/ALN.0000000000002638. PMID 30844949
- [Background] Zhu C, Yao JW, An LX, Bai YF, Li WJ. Effects of intraoperative individualized PEEP on postoperative atelectasis in obese patients: study protocol for a prospective randomized controlled trial. Trials. 2020 Jul 6;21(1):618. doi: 10.1186/s13063-020-04565-y. PMID 32631414
- [Result] Eichler L, Truskowska K, Dupree A, Busch P, Goetz AE, Zollner C. Intraoperative Ventilation of Morbidly Obese Patients Guided by Transpulmonary Pressure. Obes Surg. 2018 Jan;28(1):122-129. doi: 10.1007/s11695-017-2794-3. PMID 28707173
- [Result] Lutfi MF. The physiological basis and clinical significance of lung volume measurements. Multidiscip Respir Med. 2017 Feb 9;12:3. doi: 10.1186/s40248-017-0084-5. eCollection 2017. PMID 28194273
- [Result] Moon TS, Tai K, Kim A, Gonzales MX, Lu R, Pak T, Smith K, Chen JL, Minhajuddin AT, Nnamani N, Fox PE, Ogunnaike B. Apneic Oxygenation During Prolonged Laryngoscopy in Obese Patients: a Randomized, Double-Blinded, Controlled Trial of Nasal Cannula Oxygen Administration. Obes Surg. 2019 Dec;29(12):3992-3999. doi: 10.1007/s11695-019-04077-y. PMID 31317460
- [Result] Simon P, Girrbach F, Petroff D, Schliewe N, Hempel G, Lange M, Bluth T, Gama de Abreu M, Beda A, Schultz MJ, Pelosi P, Reske AW, Wrigge H; PROBESE Investigators of the Protective Ventilation Network* and the Clinical Trial Network of the European Society of Anesthesiology. Individualized versus Fixed Positive End-expiratory Pressure for Intraoperative Mechanical Ventilation in Obese Patients: A Secondary Analysis. Anesthesiology. 2021 Jun 1;134(6):887-900. doi: 10.1097/ALN.0000000000003762. PMID 33843980
- [Result] Hassan EA, Baraka AAE. The effect of reverse Trendelenburg position versus semi-recumbent position on respiratory parameters of obese critically ill patients: A randomised controlled trial. J Clin Nurs. 2021 Apr;30(7-8):995-1002. doi: 10.1111/jocn.15645. Epub 2021 Jan 25. PMID 33432600
- [Result] Soleimanpour H, Safari S, Sanaie S, Nazari M, Alavian SM. Anesthetic Considerations in Patients Undergoing Bariatric Surgery: A Review Article. Anesth Pain Med. 2017 Jul 11;7(4):e57568. doi: 10.5812/aapm.57568. eCollection 2017 Aug. PMID 29430407
- [Result] Jonkman AH, Ranieri VM, Brochard L. Lung recruitment. Intensive Care Med. 2022 Jul;48(7):936-938. doi: 10.1007/s00134-022-06715-z. Epub 2022 May 2. No abstract available. PMID 35499759
- [Result] Gao D, Sun L, Wang N, Shi Y, Song J, Liu X, Yang Q, Su Z. Impact of 30 degrees Reserve Trendelenburg Position on Lung Function in Morbidly Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy. Front Surg. 2022 Feb 24;9:792697. doi: 10.3389/fsurg.2022.792697. eCollection 2022. PMID 35284476
- [Result] Ball L, Pelosi P. How I ventilate an obese patient. Crit Care. 2019 May 16;23(1):176. doi: 10.1186/s13054-019-2466-x. No abstract available. PMID 31097006
- [Result] Protti A, Santini A, Pennati F, Chiurazzi C, Cressoni M, Ferrari M, Iapichino GE, Carenzo L, Lanza E, Picardo G, Caironi P, Aliverti A, Cecconi M. Lung Response to a Higher Positive End-Expiratory Pressure in Mechanically Ventilated Patients With COVID-19. Chest. 2022 Apr;161(4):979-988. doi: 10.1016/j.chest.2021.10.012. Epub 2021 Oct 16. PMID 34666011
- [Result] Yilmaz H, Kazbek BK, Koksoy UC, Gul AM, Ekmekci P, Caglar GS, Tuzuner F. Hemodynamic outcome of different ventilation modes in laparoscopic surgery with exaggerated trendelenburg: a randomised controlled trial. Braz J Anesthesiol. 2022 Jan-Feb;72(1):88-94. doi: 10.1016/j.bjane.2021.04.028. Epub 2021 May 12. PMID 33991554